CLINICAL TRIAL: NCT04319458
Title: Entertainment Education for Depression in Latinx Adults: Testing Mediators and Moderators of a Culture-Centric Narrative Intervention to Promote Help-Seeking Behavior
Brief Title: Testing Mediators and Moderators of a Fotonovela for Depression to Promote Help-seeking Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Louise Dixon De Silva, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 19-000112
Record Dates: First submitted 2019-09-06; First posted 2020-03-24 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Mental Health Literacy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fotonovela (Experimental): Fotonovela mental health literacy intervention: Secret Feelings/Sentimientos Secretos
  Interventions: Behavioral: Fotonovela
- Control (Active Comparator): Control mental health literacy intervention: NIH publication - Depression: What You Need to Know
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Fotonovela — Secret Feelings/Sentimientos Secretos
  Arms: Fotonovela
Behavioral: Control — NIH Brochure: Depression: What You Need to Know
  Arms: Control

SUMMARY:
Although rates of depression are similar in Latinx populations compared to non-Latinx whites (NLW), there are significant disparities in service utilization. Mental health literacy - one's knowledge and attitudes about mental health and treatment-seeking - is a significant predictor of help-seeking behavior and likely contributes to mental health disparities among Latinx. Understanding ways to improve mental health literacy in Latinx populations is important to reducing these disparities. Health literacy interventions that are engaging, dramatic, and culturally-relevant, such as fotonovelas (graphic novels designed to change health-related knowledge and attitudes), show promise in changing mental health literacy in Latinx populations. However, little is known about how these interventions work and for whom they are most effective. Furthermore, although there is some evidence that fotonovelas can change mental health attitudes and intent to seek treatment, their impact on help-seeking behavior is less understood. The purpose of this study is to examine 1) if narrative and cultural elements of a fotonovela for Latinx with depression (i.e., transportation, identification, and social proliferation) are important mediators in changing mental health attitudes and help-seeking behaviors and 2) if factors such as rurality, acculturation, depression severity and logistic barriers to treatment moderate these relationships.

DETAILED DESCRIPTION:
Latinx adults with depression are a particularly vulnerable population; although Latinx exhibit similar rates of depression to other racial/ethnic groups, they are less likely to seek treatment, are more likely to drop out of treatment, and thus experience greater chronicity of depression. This health disparity is likely due to a complex network of factors, but mental health literacy is one important contributing factor. Latinx are more likely to exhibit lower mental health literacy (including misconceptions, stigma, knowledge of treatment, etc.), which contributes to lower rates of treatment-seeking. Understanding how to engage Latinx in depression treatment by overcoming health literacy barriers is important in reducing health disparities.

Entertainment-education interventions are those that use popular media to engage consumers and deliver health messages. These interventions hypothesized to be useful in targeting populations with health disparities in encouraging changes in health-related behavior through dramatic and culturally-relevant narrative elements. However, no study has tested these theorized mechanisms in helping to explain changes in health literacy and subsequent health behavior.

This study will test the impact of a graphic novel about depression specifically for Latinx adults with depressive symptoms on theorized mediators, including transportation (feeling emotionally engaged in the narrative), identification (cultural relevance of characters, their language, and their appearance), and social proliferation (sharing of health information and mutual reinforcement of health behaviors). Furthermore, this study will test if these mediators help explain changes in mental health literacy and subsequent health behavior. Lastly, this study will test moderators of changes in mental health literacy and behavior to determine for whom the fotonovela has the largest impact.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* fluent in English or Spanish
* mild, moderate, or severe levels of depression
* identify as Latinx or Hispanic

Exclusion Criteria:

* receipt of psychotherapy or pharmacotherapy for mental health problems in the last 6 months
* unable to read in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Help-Seeking Behavior | 3 months
  The measure of help-seeking behavior is a checklist of behaviors that has been modified from the Service Assessment for Children and Adolescents. The measure assesses different sources of treatment, including psychiatrist, psychologist, social worker, spiritual advisors, ER visits, and traditional healers. Participants are asked if in the past 3 months, they have sought services from any of these professionals. Each item is binary (i.e., Yes or No). The total score will be calculated by summing the number of "yes" answers (i.e., the number of services used).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No